CLINICAL TRIAL: NCT07159802
Title: Restoring Lost Pink Triangle by Comparing Three Different Papillary Reconstruction Modalities: A Randomized Clinical Trial
Brief Title: Papillary Reconstruction Using Three Different Modalities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tasneem Ehab Gamal, Clinical Demonstrator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A02010250M
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-01

CONDITIONS: Papillary Reconstruction
Keywords: Papillary reconstruction; Hyalouronic acid; PRF

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hyaluronic acid group (Experimental): * The needle of the injectable HA is inserted at a 45 angle in an area 3 to 4 mm apical to the interdental papilla tip.
  * A one-point injection technique is performed on the connective tissue of the interdental papilla, ensuring the bevel is up by pointing the slant of the needle upward.
  * The amount of injection for every session is about 0.2 ml.
  * Then, the interdental papilla tip is lightly molded in the direction of the incisal edge with gauze for 1 min.
  * This procedure can be repeated up to five times during 3-week intervals until no black triangle is clinically observable (5).
  Interventions: Procedure: Papillary reconstruction
- Alb PRF group (Experimental): * A total of 9 mL of whole blood from each patient will be collected in a plastic tube.
  * It will be centrifuged at 700 g for 8 minutes at room temperature.
  * After centrifugation, the upper 2 mL of PPP will be collected in a syringe and heated for 10 minutes at 75°C to prepare denatured albumin (albumin gel).
  * Then, the tube will be given another 10 minutes to cool to room temperature.
  * The residual cells and growth factors in the buffy coat (liquid PRF) will be mixed with the cooled albumin gel and Alb-PRF gel will be ready for injection via a sterile syringe-to-syringe connector.
  * Alb-PRF gel will be injected into the papilla at a distance of 3-4 mm apical to the tip of the papilla and at an angle of 45º to the longitudinal axis of the adjacent teeth.
  * Patients will be recalled three weeks after injection to receive a booster dose (15).
  Interventions: Procedure: Papillary reconstruction
- Modified Beagle's technique group: (Experimental): * Two parallel vertical incisions are placed in the interdental gingiva starting from the coronal end of the papilla near the proximal contact points and extended apically longer than the length of the black triangle.
  * These two incisions are joined by a horizontal incision to create a pouch.
  * A partial thickness flap is raised from the apical end and gently advanced coronally towards the contact point.
  * The partial thickness is then rolled and folded on itself and sutured using 3-0 silk suture to keep it in the designated position.
  * During suturing, the suture is circumferentially wound around adjacent teeth to avoid any displacement.
  * Periodontal dressing will be given to provide mechanical protection(19).
  Interventions: Procedure: Papillary reconstruction

INTERVENTIONS:
Procedure: Papillary reconstruction — This study will be conducted to compare the effectiveness of three papillary reconstruction techniques: modified Beagle's technique, injection of albumin PRF, and injection of Hyaluronic Acid filler.
  Primary outcome: volumetric assessment of papilla regeneration. Secondary outcome: improvement of pink esthetic score.

SUMMARY:
papillary reconstruction will be done by three techniques : injection of hyaluronic acid in the base of the papilla and booster doses can be required , injection of ALB-PRF which resorbs slowly and so longer effect the last technique is minimal invasive surgery which is a modification of beagle's technique

DETAILED DESCRIPTION:
Interdental papilla (IDP) is the component of gingiva which occupies the cervical embrasure between proximal surfaces of the teeth. It is triangular when observed two dimensionally and pyramidal when viewed three dimensionally. Its shape, position, and presence are dependent upon the presence of underlying alveolar bone proper, proximal contact points, and area of adjacent teeth (1). This entity is also known as the interdental papillary house by Gonzalez et al (2), where the dimensions of the roof, floor and lateral walls of the interdental house help in maintaining the interdental papilla.

The function of the IDP is not only deflection of food debris but also acts as a barrier to protect the underlying periodontal tissues. A 'round cell infiltration' is found in the interdental papillae. The inflammatory infiltrate demonstrates a defense mechanism to the constant threat of bacterial invasion from dental plaque accumulation. The presence of the IDP also plays an essential role in aesthetics (3). The gingival unit is one of the key factors in maintaining esthetics and for this reason the presence of a normal sized and harmonically shaped IDP becomes crucial (4). It creates visual harmony between the gingiva topography and surrounding gingiva contours (5). Its deficiency can lead to a negative impact in the oral health-related quality of life and self-esteem for the patient.

If there is any defect of alveolar bone proper or adjacent tooth contact, the IPD will fail to sustain its original form resulting in empty space between teeth. This space is commonly referred as a black triangle or open gingival embrasure as a result of deficiency or loss of papilla beneath the contact points. This black triangle has many negative consequences as unpleasant appearance while smiling, food impaction and phonetic problems (6). Numerous risk factors lead to the development of this problem (7). These factors include aging, periodontal disease, loss of height of the alveolar bone relative to the interproximal contact, length of embrasure area, root angulations, tooth loss, faulty oral hygiene procedures, interproximal contact position, and triangular-shaped crowns (8, 9).

Due to its aesthetic impact and mandatory role, dentists always in a continuous challenge to restore the lost pink triangle because this region is characteristically narrow making surgery more difficult and limiting the blood supply to the associated soft tissue (5,10). Treatment options for papillary reconstruction could be surgical, non-surgical or ortho-restorative in nature which vary in long term success rates.

Currently the standard procedures for papillary reconstruction (PR) are sulcular releasing incisions, coronal flap movement and connective tissue graft (CTG) being replaced interproximally. Connective tissue graft with a coronally advanced flap is preferred more frequently than others. Despite its advantages, the presence of a second wound site and variable PR outcomes still leads the clinicians to search for alternatives (10).

Recently all the studies are directed toward less invasive techniques to minimize post operative discomfort, decrease number of surgical sites & improve patient satisfaction. These techniques include non-surgical injection of hyaluronic acid or platelet rich fibrin (PRF) and minor surgeries such as placement of PRF on semilunar incision or pedicle grafts as it will be described later.

Hyaluronan (HA) is a component in extracellular matrix that regulates the cells behavior, tissue environment and tissue regeneration. It has been extensively used in aesthetic products. Recently, HA has been introduced as a less invasive procedure to treat black triangle (11). The currently available injectable hyaluronic acid gels are polymers that are formulated by crosslinking hyaluronic acid produced by Streptococcus species. Injection is done on multiple sessions to ensure complete papilla regeneration (5).

Platelet rich fibrin is recommended as a supportive or alternative to CTG in periodontal surgery to benefit from its dense fibrin structure and growth factors content, that enhance wound healing and tissue formation (10). It plays a vital role in differentiation of precursor cells for regeneration of interdental papilla (12). Notably, involvement of PRF in neo angiogenesis could potentially reduce necrosis and shrinkage of the surgical flap (13, 14).

Injectable albumin platelet rich fibrin (Alb-PRF) is a recent form of PRF which overcomes limitations of previous forms such as rapid absorption. This modified biocompatible biologic product has a long degradation period that accelerates papilla regeneration by the continuous release of growth factors and increases the absorption time from two weeks to more than four months. Albumin gel is formed by heating the platelet-poor plasma (PPP) and mixed with liquid PRF to form Alb-PRF gel (15).

Modified Beagle's technique is another novel minimally invasive surgical approach for restoring lost IDP. The standard Beagle's technique includes partial thickness incision along the line angles of adjacent teeth on the palatal aspect then it's elevated and folded on the labial aspect. So our technique is a variant of Beagle's technique to achieve soft tissue augmentation of anterior interproximal space, without requiring a second surgical site. It consists of a small pedicle flap elevated from labial side and folded upon itself. Furthermore, this procedure is less time-consuming and surgically more simple (7).

For all methods to be successful, surgical procedures must maintain the integrity of interproximal tissues (16). Currently there are no randomized clinical trials comparing these minimal invasive methods and that's what we will explore in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 20 to 50 years. 2. Class 1 and 2 inter dental papilla loss according to Nordland & Tarnow classification (17).

  3. Adequate attached gingiva (minimum 3 mm). 4. Stage 1or 2 periodontitis (18).

Exclusion Criteria:

* 1. Smokers. 2. Chronic systemic diseases. 3. Drug usage. 4. High frenum attachment. 5. Diastema. 6. Pregnancy and lactation. 7. Stage 3 & 4 periodontitis (18). 8. Noncompliance with oral hygiene measures.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
volumetric assessment of papilla regeneration. | 6 months
  By intraoral scanner & image analysis

SECONDARY OUTCOMES:
improvement of pink esthetic score. | 6 months
  Using pink esthetic score scale

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem E Abdallah, BDS, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No